CLINICAL TRIAL: NCT03382665
Title: Prospective, Multi - Centre Clinical Evaluation of the Performance and Safety of the HYPERION Hip Endoprosthesis System in Defect Reconstruction
Brief Title: Post-market Surveillance Study With the HYPERION Hip Endoprosthesis System in Defect Reconstruction
Status: Terminated | Type: Observational
Why Stopped: CE mark will not be renewed, PMCF data no longer required
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BMETEU.CR.EU79.10
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Functional Deformities; Pseudoarthrosis; Revision of Endoprosthesis-treated Hips; Fracture, Proximal Humeral; Provision of Non-endoprosthetic Previous Operations of the Hip Joint (e.g., Transposition Osteotomies); Femur Fracture; Pseudarthrosis; Trochanteric Fractures; Bridging of Large Bone Defects; Revisions
Keywords: Revision total hip arthroplasty; Medical Device; Post Market Surveillance Study; Primary total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Pseudarthrosis; Shoulder Fractures; Femoral Fractures; Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study is a multi-center, prospective, non-controlled, consecutive cohort post market surveillance study. The objective of this study is to obtain survival and clinical outcome data on the Hyperion® system in primary and revision total hip arthroplasty.

DETAILED DESCRIPTION:
This multi-center, prospective, non-controlled, consecutive cohort post market surveillance study will serve the purpose of confirming long-term safety and performance of the Hyperion® system. The performance of the Hyperion® THA System will be evaluated using standard scoring systems (Merle d'Aubigné Score, HOOS Score). Safety will be evaluated by adverse event reporting.

The study will be performed at 6 sites, enrolling in total 70 patients. Follow-up visits are planned after 3 to 6 month, 1, 2 and 5 years. The scores will be filled in pre-operatively and post-operatively until 5 years. In order to obtain mid- to long-term patient satisfaction data the patient questionnaire will be send to the patient at 7 and 10 years, additionally. Xrays will be done pre-operatively, immediate post-operatively and at each of the Follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Patient age at least 18 years
* Fully conscious and capable patients
* Signed informed consent
* Stationary treatment
* Merle d'Aubigné < 12 Points, WOMAC Score > 25 Points
* Patients with at least one of the following indications:

Indications for primary hip replacement:

* Non-inflammatory diseases of the joints such as osteoarthritis and avascular necrosis (head necrosis)
* Rheumatoid arthritis
* Functional deformities
* Provision of non-endoprosthetic previous operations of the hip joint (e.g., transposition osteotomies)
* Treatment of pseudarthrosis, femoral neck and trochanter fractures, as well as fractures of the proximal femur affecting the head, which can not be treated by other techniques

Revision THA:

* Revision of endoprosthesis-treated hips as a result of septic or aseptic loosening, sub- and periprosthetic fractures or material failure (eg fracture of the prosthesis)
* Bridging of large bone defects (precondition: suitable proximal bone situation for a stable anchorage), i.e. for tumors

Exclusion Criteria:

* Infections
* Patients under 18 years
* Pregnant or breastfeeding patients
* Known alcohol abuse (at least 20 g alcohol per day for women and at least 40 g per day for men) or drug abuse
* Legal incapacity or restricted capacity
* Participation in another clinical trial within the last 30 days or planned participation in another clinical trial within the next 3 months
* Patients who are unable to attend to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Because of the studiesindications it is assumed that patients have a relatively high (> 60 Jahre) age at the time of their operations. Therefore a higher letality and a higher drop-out-rate is expected compared to study populations of primary hip replacement. To reach the necessery power for this clinical study at least 70 patients should be recruited.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Vivoda, Study Director — Zimmer Biomet
Locations (3):
- Germany (3):
  - Helios Klinik Hildesheim, Hildesheim
  - Klinikum Osnabrück GmbH, Osnabrück
  - Asklepios Orthopädische Klinik Lindenlohe, Schwandorf in Bayern

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients, Suffering From Severe Hip Pain and Disability: Patients in need of a total hip arthroplasty
Period: Overall Study
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability
Started (signed the informed consent) | 70
Actual Enrollment (11 patients were excluded from the study for different reasons) | 59
5 Year Follow up | 25
Completed (= longest FUP (Study completion was never reached since the study was terminated earlier).) | 25
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data available for 57 Patients
  years
    number analyzed (Participants) | 57
    (all) | 72.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 61
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI available for 56 patients
  kg/m^2
    number analyzed (Participants) | 56
    (all) | 28.9 (5.5)
Operative Side [Count of Participants; unit: Participants] — Population: Data on operative side available for 59 patients
  Participants
    number analyzed (Participants) | 59
    LEFT | 28
    RIGHT | 31

OUTCOME MEASURES:

1. Primary Outcome: Pain and Walking Ability Determined by a Merle d' Aubigné Score Increase of >4 Points.
Description: Pain and walking ability determined by a Merle d' Aubigné Score (MdA) increase of >4 points compared to the pre-operative score points.
  The patients were evaluated by the Merle d'Aubigné hip score, which evaluates pain, gait and mobility, on a scale of 1 to 6 for each item, where 1 indicates the worst and 6, the best state of the patient. The value of each item is summed to a total score. The total minimum score reached is 3, and the maximum is 18. Higher scores mean a better outcome.
Time Frame: baseline/Pre-op and 2 years (+/- 2 months)
Population: MdA score not available for all participants
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients, Suffering From Severe Hip Pain and Disability: Preop MdA scores
- Patients, Suffering From Severe Hip Pain and Disability 1: 2-year MdA scores
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability | Patients, Suffering From Severe Hip Pain and Disability 1
Number analyzed (Participants) | 54 | 35
score on a scale | 6.3 (3.7) | 13.8 (2.8)

2. Primary Outcome: Implant Survival Measured by the Number of Revisions.
Description: Implant survival is measured by the number of revisions and analysed by the Kaplan Meier method.
Time Frame: 2 years (+/- 2 month)
Population: number of revisions at 2 years
Measure: Count of Units; unit: implants
Units Other Than Participants: implants
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 39
Number analyzed (implants) | 39
implants | 11

3. Primary Outcome: WOMAC Score Value Decrease at 2-years in Min. 25 Points Compared to the Pre-operative WOMAC Score Value
Description: at 2-years post op, WOMAC score (Western Ontario and McMaster Universities Arthritis Index) has to be at least 25 points lower compared to preop values
  Scale: min 0-Max 100; Higher values mean worse outcome
Time Frame: baseline/Pre-op and 2 years (+/- 2 months)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Patients, Suffering From Severe Hip Pain and Disability 1: Preop Total WOMAC scores
- Patients, Suffering From Severe Hip Pain and Disability: 2-year Total WOMAC scores
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability 1 | Patients, Suffering From Severe Hip Pain and Disability
Number analyzed (Participants) | 41 | 26
score on a scale | 66.8 (22.4) | 27.5 (20.9)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the entire duration of the study, from first surgery to last follow up at 5 years.
Arm/Group | Patients, Suffering From Severe Hip Pain and Disability
All-Cause Mortality (participants affected / at risk) | 8/70
Serious Adverse Events (participants affected / at risk) | 38/70
Other Adverse Events (participants affected / at risk) | 33/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients, Suffering From Severe Hip Pain and Disability (N=70)
General SAE (General disorders) | 38 (38) — Serious Adverse Events were monitored/assessed without regard to the specific Adverse Event Term
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients, Suffering From Severe Hip Pain and Disability (N=70)
General AE (General disorders) | 33 (33) — Adverse Events were monitored/assessed without regard to the specific Adverse Event Term

LIMITATIONS AND CAVEATS:
Early termination of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-04): https://cdn.clinicaltrials.gov/large-docs/65/NCT03382665/Prot_SAP_000.pdf